CLINICAL TRIAL: NCT04389333
Title: Feasibility of Non-contact Magnetically-controlled Capsule Endoscopy During COVID-19 Pandemic: a Prospective, Open-label, Pilot, Randomized Trial
Brief Title: Feasibility of Non-contact Magnetically-controlled Capsule Endoscopy During COVID-19 Pandemic
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Changhai Hospital (Other)
Responsible Party: Principal Investigator, Zhuan Liao, Principal Investigator, Changhai Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: nc-MCE pilotRCT
Record Dates: First submitted 2020-05-09; First posted 2020-05-15 (Actual); Results first posted 2022-01-04 (Actual); Last update posted 2022-01-05 (Actual); Status verified 2021-12

CONDITIONS: Gastrointestinal Disease; Infectious Disease; Capsule Endoscopy
MeSH Terms: conditions — Gastrointestinal Diseases; Communicable Diseases | interventions — Endoscopy

STUDY DESIGN:
Intervention Model Description: The investigators recruited 40 patients who have related symptom and healthy people mainly from outpatient clinic or hostipal health examination center. After fully understanding the procedure of nc-MCE，patients with informed consent were randomly divided into MCE group and nc-MCE group(1:1) by using a stratified block randomization(block size four)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Non-contact MCE examination (Experimental): After an overnight fasting and drinking 1000 mL water and simethicone for gastric dilatation and preparation, the study subject positions himself (herself) on the examination bed in Room A, while the operating doctor sits in Room B at the remote control workstation instructing her to swallow the capsule via the audio-visual exchange system. After the capsule entering the stomach, the doctor manipulated the two joysticks on the remote control workstation, mobilizing the robotic magnetic arm, and simultaneously driving the precise movement and rotation of the capsule to perform the gastric examination. In order to simplify the examination procedure, the data recorder was put on the examination bed. The patient lay down after swallowing the capsule under the remote guidance of the endoscopist.
  Interventions: Device: non-contact magnetically-controlled capsule endoscopy
- MCE examination (Active Comparator): After an overnight fasting and drinking 1000 mL water and simethicone for gastric dilatation and preparation, the subjects put on the data recorder with the help of an endoscopist. Then, the endoscopist activated the capsule with the capsule locator. The patient was instructed to assume the supine or left lateral decubitus position and to swallow the capsule with a small amount of water to effectively observe the esophagus and dentate line. Then, under the guidance of the endoscopist face to face, the subject turned over on the bed to complete the examination.
  Interventions: Device: non-contact magnetically-controlled capsule endoscopy

INTERVENTIONS:
Device: non-contact magnetically-controlled capsule endoscopy — The novel non-contact magnetically-controlled capsule endoscopy (MCE) system (Ankon Technologies, Wuhan, China) (Figure 1) added a remote control workstation and an audio-visual exchange system to the original well-establish MCE system, which consisted of a robotic magnetic arm, a workstation (currently bypassed) and a capsule endoscope.

SUMMARY:
In December 2019, an outbreak of pneumonia associated with a novel coronavirus named as severe acute respiratory syndrome coronavirus 2 (SARSCoV-2) was reported in Wuhan city, China, and spread exponentially throughout China and other countries in the following weeks.

It is recommended that elective endoscopies should be deferred during the COVID-19 outbreak for the potential transmission between patients and medical staff in the statements of Asian Pacific Society for Digestive Endoscopy (APSDE-COVID statements). Therefore, exploring an alternative for patients with the requirements of endoscopy during the outbreak is of great importance.

Herein,the investigators developed an novel non-contact magnetically-controlled capsule endoscopy (Nc-MCE) system (Figure 1) adds a remote control workstation and a audio-visual exchange system to the original well-established MCE system.

This study was a open-label, prospective, randomized controlled study approved by the institutional review board of Shanghai Changhai Hospital. It was designed to evaluate the diagnostic utility, safety, feasibility and patients acceptability of Nc-MCE in patients with an indication of endoscopy, and comparing it with the result of MCE.

DETAILED DESCRIPTION:
The nc-MCE system added a remote control workstation and an audio-visual exchange system to the original well-establish MCE system.Conventional protective measures could be adopted to endoscopist. Although the endoscopist and the patient are in different rooms, the endoscopist was able to see the patient and communicate with him or her through the audio-visual exchange system all the time. In order to simplify the examination procedure, the data recorder was putted on the examination bed. The patient lay down after swallowing the capsule under the remote guidance of the endoscopist.And the endoscopist of MCE and nc-MCE was the same one with experience of more than 1000 cases of MCCG operation.

The investigators recruited 40 patients who have related symptom and healthy people mainly from outpatient clinic or hospital health examination center. After fully understanding the procedure of nc-MCE, patients with informed consent were randomly divided into MCE group and nc-MCE group(1:1) by using a stratified block randomization(block size four).

The basic characteristics of the enrolled patients were prospectively collected. The primary endpoint was the maneuverability score evaluated by endoscopist. And the investigators choose the gastric examination time,the comfort and acceptability of patients, diagnostic yield and completeness of gastric examination as the secondary endpoint. The safety endpoint of nc-MCE was evaluated by the occurrence of adverse events.

ELIGIBILITY:
Inclusion Criteria:

Signed the informed consents before joining this study

Exclusion Criteria:

(1) dysphagia or symptoms of gastric outlet obstruction, suspected or known intestinal stenosis,overt gastrointestinal bleeding,fistulas and strictures; (2)history of upper gastrointestinal surgery or suspected delayed gastric emptying; (3) Patients with poor general condition,asthma or claus trophobia; (4) Implanted metallic devices such as pacemakers,defibrillators, artificial heart valves or joint prostheses; (5) Pregnancy or mentally ill person; (6) currently participating in another clinical study;(7)communication obstacles persons.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-03-26 (Actual); Primary Completion 2020-04-26 (Actual); Study Completion 2020-05-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Zhuan Liao, MD, Study Chair — Department of Gastroenterology, Changhai Hospital, the Naval Medical University
Locations (1):
- Changhai Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chen YZ, Pan J, Luo YY, Jiang X, Zou WB, Qian YY, Zhou W, Liu X, Li ZS, Liao Z. Detachable string magnetically controlled capsule endoscopy for complete viewing of the esophagus and stomach. Endoscopy. 2019 Apr;51(4):360-364. doi: 10.1055/a-0856-6845. Epub 2019 Mar 1. PMID 30822803
- [Background] Jiang X, Pan J, Li ZS, Liao Z. Standardized examination procedure of magnetically controlled capsule endoscopy. VideoGIE. 2019 May 30;4(6):239-243. doi: 10.1016/j.vgie.2019.03.003. eCollection 2019 Jun. No abstract available. PMID 31194028
- [Background] Chiu PWY, Ng SC, Inoue H, Reddy DN, Ling Hu E, Cho JY, Ho LK, Hewett DG, Chiu HM, Rerknimitr R, Wang HP, Ho SH, Seo DW, Goh KL, Tajiri H, Kitano S, Chan FKL. Practice of endoscopy during COVID-19 pandemic: position statements of the Asian Pacific Society for Digestive Endoscopy (APSDE-COVID statements). Gut. 2020 Jun;69(6):991-996. doi: 10.1136/gutjnl-2020-321185. Epub 2020 Apr 2. PMID 32241897
- [Background] Eldridge SM, Chan CL, Campbell MJ, Bond CM, Hopewell S, Thabane L, Lancaster GA; PAFS consensus group. CONSORT 2010 statement: extension to randomised pilot and feasibility trials. Pilot Feasibility Stud. 2016 Oct 21;2:64. doi: 10.1186/s40814-016-0105-8. eCollection 2016. PMID 27965879
- [Background] Jiang B, Qian YY, Pan J, Jiang X, Wang YC, Zhu JH, Zou WB, Zhou W, Li ZS, Liao Z. Second-generation magnetically controlled capsule gastroscopy with improved image resolution and frame rate: a randomized controlled clinical trial (with video). Gastrointest Endosc. 2020 Jun;91(6):1379-1387. doi: 10.1016/j.gie.2020.01.027. Epub 2020 Jan 22. PMID 31981648

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Non-contact MCE Examination | MCE Examination
Started | 20 (From March 26th to April 26th, 2020, 20 patients were enrolled and underwent non-contract MCE in Changhai hpospital and the first medical center of PLA general hospital.) | 20 (From March 26th to April 26th, 2020, 20 patients were enrolled and accept MCE in Changhai hpospital and the first medical center of PLA general hospital.)
Completed | 20 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: From March 26, 2020 to April 26, 2020, 40 patients (19 men and 21 women) were enrolled and included in the analysis. Of them, 20 accepted MCE and 20 underwent ncMCE according to the random number table.
Groups:
- ncMCE Group: The ncMCE system adds a remote control workstation and an audio-visual exchange system to the original well-established MCE system, which was developed and tested at our medical center [10]. To simplify the preparation process, we embedded the data recorder in the examination bed. The ncMCE system separates endoscopists and patients in two rooms (control room for the endoscopist and examination room for patients), offering physical isolation for noninvasive gastric examination during the pandemic.
- MCE Group: The MCE system (Ankon Technologies Co., Ltd. Shanghai, China) consists of a guidance C-arm magnet robot, a computer workstation with ESNavi software, endoscopic capsule, capsule locator, and a vest-like data recorder that can receive capsule signals from both sides.
- Total: Total of all reporting groups
Arm/Group | ncMCE Group | MCE Group | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.1 (14.8) | 53.5 (9.2) | 49.8 (12.72)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 12 | 21
  Male | 11 | 8 | 19
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 20 | 20 | 40
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
History of abdominal surgery [Count of Participants; unit: Participants] | 4 | 6 | 10
Diabetes [Count of Participants; unit: Participants] | 2 | 1 | 3
Smoking history [Count of Participants; unit: Participants] | 3 | 6 | 9
Drinking history [Count of Participants; unit: Participants] | 6 | 7 | 13
Indication:Symptoms [Count of Participants; unit: Participants] | 18 | 14 | 32
Indication:Health checkup [Count of Participants; unit: Participants] | 2 | 6 | 8
Indication:Abdominal pain [Count of Participants; unit: Participants] | 9 | 3 | 12
Indication:Abdominal distension [Count of Participants; unit: Participants] | 7 | 6 | 13
Indication: Acid reflux [Count of Participants; unit: Participants] | 0 | 2 | 2
Indication: Others [Count of Participants; unit: Participants] — The other indications included other inspection reasons except for abdominal pain, abdominal distension, acid reflux and health checkup.
  Participants | 0 | 3 | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Complete Observation
Description: The number of participants with complete observation. Complete observation of the mucosa means over 90% of the mucosa observed in gastric cardia, fundus, body, angulus, antrum and pylorus.
Time Frame: During the procedure
Measure: Count of Participants; unit: Participants
Arm/Group | ncMCE Group | MCE Group
Number analyzed (Participants) | 20 | 20
Participants | 20 | 20

2. Secondary Outcome: Maneuverability Score
Description: Maneuverability score was the sum of four subjective scores rated by the operator (signal transmission quality score, operating comfort score, gastric visualization score and study subject compliance score), each of which ranged from 1 to 5 denoting the lowest to the highest degree of satisfaction and the range of total score from 0 to 20. The higher the score, the better the maneuverability.
Time Frame: During the procedure
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | ncMCE Group | MCE Group
Number analyzed (Participants) | 20 | 20
score on a scale
  Transmission quality | 4.5 [4.5 to 5] | 5 [5 to 5]
  Comfortableness | 5 [5 to 5] | 5 [5 to 5]
  Visualization | 5 [5 to 5] | 5 [4 to 5]
  Compliance of patients | 5 [5 to 5] | 5 [5 to 5]
  Total | 19.25 [18.63 to 20] | 20 [19 to 20]

3. Secondary Outcome: Gastric Examination Time(GET)
Description: GET was defined as the time taken for the endoscopist to complete the gastric examination to his or her satisfaction
Time Frame: During the procedure
Measure: Mean (Inter-Quartile Range); unit: minute
Arm/Group | ncMCE Group | MCE Group
Number analyzed (Participants) | 20 | 20
minute | 12.3 [7.5 to 16.3] | 7.2 [6.5 to 8.9]

4. Secondary Outcome: the Comfort and Acceptability of Patients
Description: The investigators use a satisfaction questionnaire to evaluate the comfort and acceptability of each patient by two sub questionnaires, which was pre-procedure patient perception (3 items, ranged from 0 to 12 ) and post-procedure patient satisfaction (12 items, ranged from 0 to 48) .The higher the score, the worse the patient's satisfaction.
Time Frame: After the procedure(within 5 days)
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | ncMCE Group | MCE Group
Number analyzed (Participants) | 20 | 20
score on a scale
  Pre-procedure patient perception | 9 [8 to 9] | 9 [8 to 9]
  Post-procedure patient satisfaction | 45 [42.3 to 46.8] | 44 [42 to 45]

5. Secondary Outcome: The Total Number of Patients Who Who Had a Diagnosis of Positive Findings
Description: It was calculated using the following formula: number of patients with positive findings divided by the total number of patients that underwent examination.
Time Frame: after the procedure(within 5 days)
Measure: Count of Participants; unit: Participants
Groups:
- ncMCE Group: The ncMCE system adds a remote control workstation and an audio-visual exchange system to the original well-established MCE system, which was developed and tested at our medical center. To simplify the preparation process, we embedded the data recorder in the examination bed. The ncMCE system separates endoscopists and patients in two rooms (control room for the endoscopist and examination room for patients), offering physical isolation for noninvasive gastric examination during the pandemic.
Arm/Group | ncMCE Group | MCE Group
Number analyzed (Participants) | 20 | 20
Participants
  Polyp | 2 | 3
  Erosion | 2 | 1
  Ulcer | 0 | 2
  Total | 4 | 6

6. Other Pre Specified Outcome: Adverse Events
Description: Each patient was followed up for 2 weeks by telephone and hospital information system to confirm capsule excretion and any adverse events (AEs), including COVID-19 infection.
Time Frame: During and within 2 weeks after the procedure
Population: Each patient was followed up for 2 weeks by telephone and hospital information system to confirm capsule excretion and any adverse events (AEs), including COVID-19 infection.
Measure: Count of Participants; unit: Participants
Arm/Group | ncMCE Group | MCE Group
Number analyzed (Participants) | 20 | 20
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: safety based on the occurrence of adverse events (AEs) including infection which was recorded till the 14 days after swallowing the capsule.
Description: Each patient was followed up for 2 weeks by telephone and hospital information system to confirm capsule excretion and any adverse events (AEs), Possible adverse events included capsule retention, dysphagia, capsule incarceration, infection of SARS-COV-2.
Arm/Group | ncMCE Group | MCE Group
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-02-03): https://cdn.clinicaltrials.gov/large-docs/33/NCT04389333/Prot_SAP_000.pdf